CLINICAL TRIAL: NCT04706208
Title: Identifying Body Awareness-related Brain Network Changes During Cognitive Multisensory Rehabilitation for Reduced Neuropathic Pain in People With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMR-2020-29297
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One time testing - able-bodied healthy adults (Other): Participants in this arm will be able-bodied healthy adults who will not receive an intervention.
  This is just a one time testing of clinical assessments (over zoom), one MRI scan, and an optional blood draw test.
  Interventions: Behavioral: Clinical Assessment; Behavioral: Magnetic Resonance Imaging (MRI); Other: OPTIONAL: blood draw
- Usual Care, then Cognitive Multisensory Therapy - adults with spinal cord injury + neuropathic pain. (Experimental): This is a delayed treatment arm phase I randomized controlled trial (RCT) for participants with spinal cord injury and neuropathic pain. Participants in this arm will first receive usual care and then switch over to the experimental cognitive multisensory therapy training.
  Interventions: Behavioral: Cognitive Multisensory Therapy; Other: Usual Care; Behavioral: Clinical Assessment; Behavioral: Magnetic Resonance Imaging (MRI); Other: OPTIONAL: blood draw
- Cognitive Multisensory Therapy, then Usual Care - adults with spinal cord injury + neuropathic pain. (Experimental): This is a delayed treatment arm phase I randomized controlled trial (RCT) for participants with spinal cord injury and neuropathic pain. Participants in this arm will first receive the experimental cognitive multisensory therapy training and then switch over to usual care.
  Interventions: Behavioral: Cognitive Multisensory Therapy; Other: Usual Care; Behavioral: Clinical Assessment; Behavioral: Magnetic Resonance Imaging (MRI); Other: OPTIONAL: blood draw

INTERVENTIONS:
Behavioral: Cognitive Multisensory Therapy — Cognitive multisensory rehabilitation (CMR) is a type of physical therapy that incorporates conscious perception of body positions and movements during (multi)sensory discrimination exercises. The treating therapists will give 40 minutes of discrimination exercises embedded in functional movements followed by 5 minutes of applying the learned strategies during activities of daily living. CMR uses several types of discrimination exercises: Participants discriminated shapes, length, weight, distance, resistance, textures or compare kinesthetic information with visual information for integration of multisensory information. Solving the discrimination task is combined with reflection and a learning process, prompted by the therapist on how the limb (was) moved or was positioned.
  Arms: Cognitive Multisensory Therapy, then Usual Care - adults with spinal cord injury + neuropathic pain.; Usual Care, then Cognitive Multisensory Therapy - adults with spinal cord injury + neuropathic pain.
Other: Usual Care — Standard of care treatment for neuropathic pain after spinal cord injury
  Arms: Cognitive Multisensory Therapy, then Usual Care - adults with spinal cord injury + neuropathic pain.; Usual Care, then Cognitive Multisensory Therapy - adults with spinal cord injury + neuropathic pain.
Behavioral: Clinical Assessment — Clinical assessments are detailed below. Screening will include demographic and general health data; mini mental state evaluation (MMSE)-short version; Edinburgh handedness inventory; and the kinesthetic and visual imagery questionnaire (KVIQ).
Behavioral: Magnetic Resonance Imaging (MRI) — The MRI scanning will include structural scans, resting-state functional MRI, and 4 task-based functional MRI.
Other: OPTIONAL: blood draw — This part is OPTIONAL: 38ml of blood will be taken one time (for able body adults) or at 3 time points (for adults with spinal cord injury and neuropathic pain.

SUMMARY:
Many adults with spinal cord injury (SCI) suffer from long-term debilitating neuropathic pain. Available treatments, including opioids, are ineffective at eliminating this pain. Based on preliminary data from Dr Morse and from Dr Van de Winckel, we have demonstrated that brain areas that are important for body awareness and pain perception (parietal operculum, insula) have weaker brain connectivity in adults with spinal cord injury than in able-bodied healthy adults and that Cognitive Multisensory Rehabilitation (CMR) can restore these networks. This study uses a delayed treatment arm phase I randomized controlled trial (RCT) for adults with SCI and a comparison of baseline outcomes in adults with SCI vs able-bodied healthy adults to address two aims:

AIM 1: Determine baseline differences in resting-state and task-based fMRI activation and connectivity in adults with SCI compared to able-bodied healthy controls.

AIM 2: Identify changes in brain activation and connectivity, as well as behavioral outcomes in pain and body awareness in adults with SCI after CMR versus standard of care.

DETAILED DESCRIPTION:
One of the reasons for the current lack of effective therapies is that underlying mechanisms of neuropathic pain after SCI are not yet fully understood. Nonetheless, as suggested by numerous studies, because of the spinal injury, the inflow of sensory information is dramatically altered. Therefore, the brain is missing sensory information or receiving incorrect sensory information, which may alter the brain circuitry related to pain sensation, which in turn may drive the perception of neuropathic pain.

Cognitive multisensory rehabilitation (CMR), developed for motor recovery after stroke, has shown to be effective for treating adults with chronic pain, i.e., after shoulder impingement when compared to traditional physical therapy; or in a case study of severe phantom limb pain after below the knee amputation, resulting in such substantial pain reduction that the patient could finally be fitted with a prosthesis and walk. CMR is thought to be effective because it restores mental body representations by recalibrating sensations in combination with a focus on body awareness. Body awareness is often impaired in people with chronic pain and with dysfunctions in the sensory and motor networks, such as after SCI.

This study uses a delayed treatment arm phase I randomized controlled trial (RCT) for adults with SCI and a comparison of baseline outcomes in adults with SCI vs able-bodied healthy adults to address two aims:

AIM 1: Determine baseline differences in resting-state and task-based fMRI activation and connectivity in adults with SCI compared to able-bodied healthy controls.

AIM 2: Identify changes in brain activation and connectivity, as well as behavioral outcomes in pain and body awareness in adults with SCI after CMR versus standard of care.

More information: https://med.umn.edu/rehabmedicine/research/sci-neuropathic-pain

ELIGIBILITY:
Inclusion Criteria:

SCI participants:

* SCI of ≥ 3months
* medically stable with paraplegia (ASIA grade A-C, who can self-transfer with some assistance)
* neuropathic pain (>3 on the numeric pain rating scale)

Able-bodied participants:

* sex and age matched
* healthy, able-bodied

Exclusion Criteria:

- MRI contra-indications (stabilizing hardware is typically MRI safe) including seizures, cognitive impairment, or other major medical complications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale (NPRS) - part of the International SCI Basic Pain Data Set | weekly during the two intervention periods (each 12 weeks)
  The numeric pain rating scale assesses the highest, lowest and average pain ratings over the past week. The 1-10 numerical pain rating scale has been recommended by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus group for use in pain clinical trials and by the 2006 National Institute on Disability and Rehabilitation Research (NIDRR) SCI Pain outcome measures consensus group. This scale is recommended to standardize pain outcomes across studies.

SECONDARY OUTCOMES:
Physical Activity Recall Questionnaire | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  This 16 item questionnaire asks about physical activity inside of the house and away from the house (including daily physical tasks) as well as hours of sleep. Time to administer: approximately 10 minutes.
Pittsburgh Sleep Quality Index (PSQI) | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  This 10-item questionnaire asks about duration and quality of sleep and reasons for not sleeping well through the night. Time to administer: approximately 6 minutes.
Spielberger State-Trait Anxiety Inventory | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  This questionnaire asks about different moods in general (trait- 19 items) and at the moment of the testing (state- 20 items). Scoring between 1-4 reflecting "almost never" to "almost always" for trait, and "not at all" to "very much so" for state)Time to administer: approximately 5 minutes.
Patient Health Questionnaire (PHQ-9) | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  The PHQ-9 is a self-report questionnaire, which assesses the presence and intensity of depressive symptoms. There are 9 items scored from 0 to 3 based on the frequency of occurrence of depression symptoms in the past two weeks, 0= not at all, 1=several days, 2=more than half the days, 3= nearly every day. Total score is a sum of all items scores and should be interpreted as follows:
  5-9 Minimal Symptoms 10-14 Moderate depression 15-20 Moderately Severe depression >20 Severe depression
  And a single question rates how difficult problems have made it to do work, take care of things at home or get along with other people, using a 4-level scale ranging from not difficult at all to externally difficult.
  Total score range: 0-27
  It takes 3 minutes to finish this questionnaire.
Moorong Self-Efficacy Scale (MSES) | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  The Moorong Self-Efficacy Scale contains 16 items rated on a 7-point Likert scale from 1 (very uncertain) to 7 (very certain). Totals score is calculated as a sum of the 16 items scores. Total scores range from 16 to 112, with higher scores reflecting high self efficacy.
WHOQOL-BREF | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  The WHOQOL- BREF assesses quality of life within the context of an individual's culture, value systems, personal goals, standards and concerns in the last two weeks. This is a self-report questionnaire 26 items assessing 4 quality domains of quality of life (QOL): physical health (7 items), psychological health (6 items), social relationships (3 items) and environmental (8 items). In addition, two other items measure overall QOL and general health.
  Items are rated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw item score. The mean score of items within each domain is used to calculate the domain score. After computed the scores, they transformed linearly to a 0-100-scale. Score of each domain is reported. A higher score indicating a higher quality of life.
Revised Body Awareness Rating Questionnaire (BARQ) | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  The Body Awareness Rating Questionnaire (BARQ) is a self-report questionnaire designed to capture how individuals with long-lasting musculoskeletal pain reflect on their own body awareness. This questionnaire contains 12 items rated on a scale from 0 (completely disagree) to 3 (completely agree). The total score is a sum of all items and ranges from 0 to 36, with lower scores indicating higher body awareness.
Tampa Scale For Kinesiophobia | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  The Tampa Scale for Kinesiophobia is a 17-item questionnaire measuring fear related to exercise and movement. Items are rated on a scale of 1 (strongly disagree) to 4 (strongly agree). A total score is calculated by summing the individual item scores after inversion of the individual scores for items 4, 8, 12 and 16. Higher scores indicated greater kinesiophobia.
Physical Activity Enjoyment Scale (PACES) | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  The Physical Activity Enjoyment Scale contains 18 items that are rated on a 7-point scale. 11 items are scored in reverse order. Total scores range from 18 to 126, with higher scores indicating greater level of enjoyment.
Patient Specific Functional Scale | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  The participants will self-identify goals related to activities in daily life that are important to them. The participants will rate them at each time point between 0 (i.e., unable to do the activity without pain) and 10 (able to do the activity without pain).This is a valid measure to assess disability in individuals with chronic pain.101 Time to administer: 5 minutes
International SCI Basic Pain Data Set | baseline - mid evaluation (after 12 weeks) - final evaluation (after second period of 12 weeks)
  Aside from NPRS (below), The International Spinal Cord Injury Pain Data Set also assesses dimensions of pain (i.e. intensity of pain, time of day, location, occurrence, etc.), and pain interference with mood, activity, and sleep. Time to administer: 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van de Winckel, Van de Winckel, Principal Investigator — University of Minnesota
Locations (1):
- University of MInnesota (Brain Body Mind Lab, Division of Physical Therapy, Department of Rehab Med, Medical School), Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets (de-identified individual participant data and data dictionary) analyzed for this study can be found in the Dryad repository and will be made available upon publication of the article.

REFERENCES:
- [Background] Van de Winckel A, Carpentier S, Deng W, Bottale S, Hendrickson T, Zhang L, Wudlick R, Linnman C, Battaglino R, Morse L. Identifying Body Awareness-Related Brain Network Changes After Cognitive Multisensory Rehabilitation for Neuropathic Pain Relief in Adults With Spinal Cord Injury: Protocol of a Phase I Randomized Controlled Trial. Top Spinal Cord Inj Rehabil. 2022 Fall;28(4):33-43. doi: 10.46292/sci22-00006. Epub 2022 Nov 15. PMID 36457363
- [Background] Van de Winckel A, Carpentier ST, Deng W, Bottale S, Zhang L, Hendrickson T, Linnman C, Lim KO, Mueller BA, Philippus A, Monden KR, Wudlick R, Battaglino R, Morse LR. Identifying Body Awareness-Related Brain Network Changes after Cognitive Multisensory Rehabilitation for Neuropathic Pain Relief in Adults with Spinal Cord Injury: Delayed Treatment arm Phase I Randomized Controlled Trial. medRxiv [Preprint]. 2023 Feb 10:2023.02.09.23285713. doi: 10.1101/2023.02.09.23285713. PMID 36798345
- See also: Brain Body Mind Lab website link for the AIRP study — https://med.umn.edu/rehabmedicine/research/sci-neuropathic-pain